CLINICAL TRIAL: NCT04061044
Title: A Prospective, Multicenter, Open Label Extension Study to Evaluate the Long Term Safety of OTX-TP
Brief Title: A Study to Evaluate the Long Term Safety of OTX-TP (Sustained Release Travoprost) Intracanalicular Insert
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-Protocol-0047
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Open Angle Glaucoma and Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Ophthalmic Insert

INTERVENTIONS:
Drug: Ophthalmic Insert — Travoprost, 0.32 mg
  Other Names: OTX-TP

SUMMARY:
To evaluate the long term safety of repeat dose OTX-TP, a sustained release travoprost drug product, placed in the canaliculus of the eyelid in the treatment of subjects with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Had prior bilateral treatment and completion, through a minimum of week 12, of the OTX-16-002 trial
* Are informed of the nature of the study and subject is able to comply with study requirements and visit schedule for one year
* Have provided written informed consent, approved by the appropriate Institutional Review Board

Exclusion Criteria:

* Had more than 1 replacement, per eye, during participation in the OTX-16-002 trial
* Had punctal or canaliculi related adverse events during the OTX-16-002 trial which required discontinuation (e.g., canaliculitis)
* Used prohibited medications during the OTX-16-002 study, or the period between OTX-16-002 and this trial (with the exception of short term medication used to treat an adverse event or rescue therapy)
* Missed more than 2 visits during participation in the OTX-16-002 trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Adverse Events (Safety and Tolerability) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- ApexEye, Cincinnati, Ohio, United States

DOCUMENTS (2):
  • Study Protocol (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT04061044/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT04061044/SAP_001.pdf